CLINICAL TRIAL: NCT01247818
Title: A Phase 2 Dose-Randomized, Vehicle-Controlled Study of PH-10-Aqueous Hydrogel for the Treatment of Plaque Psoriasis
Brief Title: Randomized Study of PH-10 for Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provectus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PH-10-PS-23
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Rose Bengal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PH-10 Treatment (High Dose Cohort) (Experimental)
  Interventions: Drug: PH-10 (0.01% Rose Bengal)
- PH-10 Treatment (Mid Dose Cohort) (Experimental)
  Interventions: Drug: PH-10 (0.005% Rose Bengal)
- PH-10 Treatment (Low Dose Cohort) (Experimental)
  Interventions: Drug: PH-10 (0.002% Rose Bengal)
- Vehicle Control (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: PH-10 (0.002% Rose Bengal) — PH-10 will be applied daily for 28 days to skin areas affected by mild to moderate psoriasis.
  Arms: PH-10 Treatment (Low Dose Cohort)
Drug: PH-10 (0.005% Rose Bengal) — PH-10 will be applied daily for 28 days to skin areas affected by mild to moderate psoriasis.
  Arms: PH-10 Treatment (Mid Dose Cohort)
Drug: PH-10 (0.01% Rose Bengal) — PH-10 will be applied daily for 28 days to skin areas affected by mild to moderate psoriasis.
  Arms: PH-10 Treatment (High Dose Cohort)
Drug: Vehicle — PH-10 vehicle will be applied daily for 28 days to skin areas affected by mild to moderate psoriasis.
  Arms: Vehicle Control

SUMMARY:
PH-10 is an aqueous hydrogel formulation of rose bengal disodium (RB) for topical administration to the skin, and is being studied for the treatment of cutaneous skin disorders, specifically psoriasis and atopic dermatitis. This multicenter phase 2 study of subjects randomized sequentially by center to one of four treatment cohorts will assess efficacy and safety of topical PH-10 applied once daily to areas of mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 or older.
* Presence of mild to moderate plaque psoriasis on the trunk or extremities (excluding palms, soles, scalp, and facial or intertriginous areas).
* Fitzpatrick skin type I-VI.
* Written informed consent by the subject or legal guardian.

Exclusion Criteria:

* Female subjects of childbearing potential who are pregnant, attempting to conceive, not using effective contraception, or who are nursing an infant.
* Subjects who have received psoralen plus ultraviolet A (PUVA) therapy or systemic antipsoriatic therapy (immunosuppressants, cytostatics, corticosteroids) within 28 days of study initiation (two weeks for methotrexate).
* Subjects who have received ultraviolet B (UVB) light therapy within 14 days of study initiation.
* Subjects who have received topical antipsoriatic therapy (including corticosteroids, tar, anthralin or Vitamin D analogs) to the study plaque areas within 14 days of study initiation.
* Subjects who have received agents posing a clinically significant risk of photosensitivity reaction within 5 half-lives of study initiation.
* Subjects who have received any approved or investigational biologic drug therapy for psoriasis within 90 days or 5 half-lives of study initiation.
* Subjects who have participated in a clinical research study within 28 days of study initiation.
* Subjects with a history of porphyria, systemic lupus erythematosus or xeroderma pigmentosum.
* Subjects with clinical conditions that, in the opinion of the Investigator may pose a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is "Treatment Success," a static endpoint assessed at Day 29 after initial PH-10 treatment and defined as 0 or 1 on all Psoriasis Severity Index (PSI) components and 0 or 1 on the Plaque Response scale. | 28 days
The primary safety endpoint is incidence of adverse experiences, including pain and dermatologic/skin toxicity (incidence, severity, frequency, duration and causality). | 8 weeks

SECONDARY OUTCOMES:
Psoriasis Severity Index (PSI) score changes at each visit from Day 1 pre-treatment. | 8 weeks
Plaque Response score changes at each visit from Day 1 pre-treatment. | 8 weeks
Pruritus Self-Assessment score changes at each visit from Day 1 pre-treatment. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wachter, Ph.D., Study Director — Provectus Pharmaceuticals
Locations (4):
- United States (4):
  - Dermatology Specialists, Inc., Oceanside, California
  - International Dermatology Research, Miami, Florida
  - Mount Sinai School of Medicine, New York, New York
  - Wake Research Associates, Raleigh, North Carolina